CLINICAL TRIAL: NCT06616909
Title: Advance Care Planning Impact on the Consistency of Older Adults With Lung Cancer and Their Potential Surrogates Regarding Life-Sustaining Treatment Preferences
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202407186RIND
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Advanced Care Planning (ACP); ELDERLY PEOPLE; Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- game ACP module (Experimental): ,Using board games as an activity intervention, a tool for discussion between elderly people with lung cancer and potential agents
  Interventions: Behavioral: ACP GAME
- ACP Manual (Placebo Comparator)
  Interventions: Behavioral: acp manual

INTERVENTIONS:
Behavioral: ACP GAME — ,Using board games as an activity intervention, a tool for discussion between elderly people with lung cancer and potential agents
  Arms: game ACP module
Behavioral: acp manual — acp manual
  Arms: ACP Manual

SUMMARY:
Background: Globally and nationally, malignant tumors persist as the leading cause of high incidence and mortality rates. In Taiwan, cancer tops the list of causes of death, with the elderly being predominantly affected, especially by lung cancer, which is the most prevalent type with the highest mortality and incidence rates in the nation. The Patient Autonomy Rights Act, implemented by the government in 2019, is designed to promote advance medical care consultation in medical institutions, respecting patient's autonomous decisions. In Chinese culture, medical decisions are typically family-oriented rather than individualistic, leading the elderly to frequently rely on their relatives'choices. This cultural practice may prevent meaningful conversations between potential agents and the elderly, causing misunderstandings of the elderly's preferences and affecting the consistency of medical decisions. Presently, interventions like board games for Advance Care Planning (ACP) are not well received, highlighting the need for more captivating content in intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. lung cancer age ≧ 60
2. The elderly with lung cancer are conscious and have no severe visual or hearing impairment.

3.3. The potential agent is designated by the elderly person with lung cancer who may be a family member who may make medical decisions in the future. The potential agent must be at least 18 years old.

Exclusion Criteria:

1. People with severe hearing loss and visual impairment who are unable to communicate in Mandarin and Taiwanese.
2. The potential agent is under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Consistency in subsistence disposal preferences between the elderly and potential agents | Outcome Measure Total (3 Time Points): First time: before intervention .Second time: 2 weeks after intervention . Last time: 6 weeks after intervention
  Life Support Preferences Questionnaire (LSPQ).

SECONDARY OUTCOMES:
STAI | Outcome Measure Total (4 Time Points): First time: Before intervention. Second time: After intervention. Third time: 2 weeks after intervention .Last time: 6 weeks after intervention
  The State-Trait Anxiety Inventory The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided